CLINICAL TRIAL: NCT07295145
Title: BeFab: An International, Multi-centre Observational Study to Evaluate Safety, Performance, and Clinical Benefit of Bentley Bridging Stent Graft Systems
Brief Title: Bentley Bridging Stent Graft Study
Acronym: BeFab
Status: Not yet recruiting | Type: Observational
Sponsor: Bentley InnoMed GmbH (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Other Study IDs: PM08-01 BeFab
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endovascular aortic repair (EVAR) — The primary goal of EVAR is to bypass the aneurysm sac with the aortic endovascular graft. Through isolation of the aneurysm sac, the blood pressure on the affected aortic tissue is reduced. This prevents aneurysm growth, which is otherwise associated with an elevated risk of rupture. As the pressure on the aneurysm sac is minimized, the current risk of rupture is also mitigated.
  In case that arteries branch off from the aorta in the area of the aneurysm, or at the proximal and distal sealing zones of the endograft, complex EVAR approaches are employed, which include stenting of the aortic branches (mostly renal and visceral arteries, also called target vessels) in addition to implantation of an aortic endovascular graft. A distinction is made between different variants of complex EVAR procedures, which comprise fenestrated endovascular aneurysm repair (FEVAR), branched endovascular aneurysm repair (BEVAR) and hybrid approaches.

SUMMARY:
This international, observational multi-centre observational study of the devices BeFlared FEVAR Stent Graft System (BeFlared), BeGraft Stent Graft System (BeGraft), and BeGraft Plus Stent Graft System (BeGraft Plus) will monitor technical success of the implantation, data regarding clinical performance, clinical benefit, as well as potential unknown side effects for the use as bridging stent grafts in combination with fenestrated aortic endovascular grafts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients having complex abdominal aortic aneurysms suitable for an endovascular repair with a fenestrated and/or branched aortic endovascular graft in combination with one Bentley bridging stent graft per reno-visceral artery in accordance with the IFU of BeFlared, BeGraft or BeGraft Plus. Use of different products for different target vessels is allowed. Use of stents from other manufacturers for other reno-visceral arteries is allowed.
* Patient is capable and willing to sign the informed consent and agrees to fulfil follow-up requirements
* Patients ≥18 years of age at the time of consent

Exclusion Criteria:

* Patients with contraindications as listed in the IFUs
* Previous stenting of the target vessel
* Extension/relining of Bentley BSGs
* Prior EVAR procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having complex abdominal aortic aneurysms
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Target vessel instability at 12 months, defined as bridging stent-specific occlusion, stenosis, endoleak Type Ic/IIIc, or re-intervention | 12 months post index procedure

SECONDARY OUTCOMES:
Target vessel instability defined as bridging stent-specific occlusion, stenosis, endoleak Type Ic/IIIc, or re-intervention | 1 month, 24 months, 36 months, 48 months, and 60 months post index procedure
Procedure-related complications | during procedure, at discharge and 1 month and 12 months post index procedure
Bridging stent-related complications | during procedure, and 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
technical success defined as correct positioning and deployment of bridging stent grafts | during procedure
Primary patency rate defined as uninterrupted patency with no occlusion | 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
Secondary patency rate | 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
Freedom from secondary procedures | 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
Freedom from bridging stent related endoleaks | 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
Post-procedure Major adverse event rate | 1 month post procedure
Freedom from aneurysm-related death | 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
Freedom from aortic aneurysm maximum diameter increase | 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
Device implantation time | during procedure
Total procedure time | during procedure
total patient radiation dose | during procedure
total time of fluoroscopy | during procedure
total volume of received contrast medium | during procedure
Patient blood loss | during the procedure
duration of ICU stay | 1 month post index procedure
duration of total hospital stay | 1 month and 12 months post index procedure
mortality rate at 30 days | 1 month post index procedure
Quality of life score | 1 month, 12 months, 24 months, 36 months, 48 months, and 60 months post index procedure
  EQ5D